CLINICAL TRIAL: NCT05735223
Title: A Prospective Study to Evaluate the Impact of Maximal Urethral Length Preservation Technique During Robotic Laparoscopic Prostatectomy in Terms of Continence Rates
Brief Title: A Prospective Study to Evaluate the Impact of Maximal Urethral Length Preservation Technique During Robotic Laparoscopic Prostatectomy on the Stretched Flaccid Penile Length and Continence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larkin Health System (Other)
Responsible Party: Principal Investigator, Balaji Reddy, MD, Principal Investigator, Larkin Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LCH-2-092019
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Prostate Adenocarcinoma; Incontinence Stress; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: In an IRB approved study, we prospectively evaluated the stretched flaccid penile length (SFPL) pre and post robot assisted laparoscopic radical prostatectomy (RALP) in subjects with a diagnosis of prostate cancer. The multiparametric MRI (MP-MRI) was utilized for surgical planning if available preoperatively. Repeated measures t-test, linear regression and 2-way ANOVA analyses were performed.
Masking Description: Stretched flaccid penile length (SFPL) was measured by a single male assessor at preoperative visit, and at the time of catheter removal (10 days post-surgery). The subjects were blinded to the measurements to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stretched flaccid penile length (SFPL) following RALP. (Experimental): Stretched flaccid penile length (SFPL) was measured by a single male assessor at preoperative visit, and at the time of catheter removal (10 days post-surgery).
  Interventions: Procedure: Maximal urethral length preservation technique of robot assisted radical prostatectomy (RALP).

INTERVENTIONS:
Procedure: Maximal urethral length preservation technique of robot assisted radical prostatectomy (RALP). — Stretched flaccid penile length (SFPL) was measured by a single male assessor at preoperative visit, and at the time of catheter removal (10 days post-surgery). The subjects were blinded to the measurements to prevent bias. Multiparametric MRI (MP-MRI) of the prostate were reviewed when available for surgical planning. All subjects underwent RALP with MULP using the technique previously published by Hamada et al. Continence defined as requiring no pads was assessed at 3 and 6 months postoperatively.

SUMMARY:
After robotic prostatectomy, besides erectile function and achievement of oncological control, staying dry is also a very important desire expressed frequently by the patients. This has led to the concept of trifecta achievement after robotic prostatectomies. Hence, continence preserving prostatectomies are the order of the day today. Patient acceptance to surgery is low if the continence cannot be assured preoperatively. Many techniques have been promulgated in the last two decades.

The investigators present a novel technique of maximal urethral length preservation during surgery as an effective method of continence preservation. The investigators hypothesize that maximal preservation of urethra would lead to improved and early continence after robotic prostatectomy. The investigators also hypothesize that urethral preservation spares penile length shortening. The investigators therefore propose to prospectively evaluate penile length shortening.

While penile length change after radical prostatectomy has been studied in the past, the investigators like to assess the penile morphometric assessment following the novel technique of maximal urethral length preservation radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria: All men undergoing robot assisted laparoscopic radical prostatectomy (RALP).

-

Exclusion Criteria:

1. Exposure to androgen deprivation therapy
2. Prior treatment for prostate cancer
3. Metastatic prostate cancer
4. History of hypospadias or urethral reconstruction
5. History of penile implant, intracorporal injections, intraurethral suppositories
6. Prior pelvic surgery. -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Penile Length | 10 days post operatively
  Stretched Flaccid Penile Length

SECONDARY OUTCOMES:
Urinary continence | 3 months and 6 months postoperatively
  Pads used.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Razdan, MD, MCh, Study Chair — Larkin Health System; Balaji Reddy, MD, Principal Investigator — Larkin Health System
Locations (1):
- Larkin Health System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frey AU, Sonksen J, Fode M. Neglected side effects after radical prostatectomy: a systematic review. J Sex Med. 2014 Feb;11(2):374-85. doi: 10.1111/jsm.12403. Epub 2013 Nov 25. PMID 24267516
- [Background] Paparel P, Akin O, Sandhu JS, Otero JR, Serio AM, Scardino PT, Hricak H, Guillonneau B. Recovery of urinary continence after radical prostatectomy: association with urethral length and urethral fibrosis measured by preoperative and postoperative endorectal magnetic resonance imaging. Eur Urol. 2009 Mar;55(3):629-37. doi: 10.1016/j.eururo.2008.08.057. Epub 2008 Sep 2. PMID 18801612
- [Background] Kadono Y, Machioka K, Nakashima K, Iijima M, Shigehara K, Nohara T, Narimoto K, Izumi K, Kitagawa Y, Konaka H, Gabata T, Mizokami A. Changes in penile length after radical prostatectomy: investigation of the underlying anatomical mechanism. BJU Int. 2017 Aug;120(2):293-299. doi: 10.1111/bju.13777. Epub 2017 Feb 8. PMID 28181381
- [Background] Hamada A, Razdan S, Etafy MH, Fagin R, Razdan S. Early return of continence in patients undergoing robot-assisted laparoscopic prostatectomy using modified maximal urethral length preservation technique. J Endourol. 2014 Aug;28(8):930-8. doi: 10.1089/end.2013.0794. Epub 2014 Apr 16. PMID 24739066
- [Background] Munding MD, Wessells HB, Dalkin BL. Pilot study of changes in stretched penile length 3 months after radical retropubic prostatectomy. Urology. 2001 Oct;58(4):567-9. doi: 10.1016/s0090-4295(01)01270-5. PMID 11597540
- [Background] Hammerer P, Huland H. [Urodynamic changes after radical prostatectomy]. Urologe A. 1997 Nov;36(6):535-9. doi: 10.1007/s001200050133. German. PMID 9487589
- [Background] Fraiman MC, Lepor H, McCullough AR. Changes in Penile Morphometrics in Men with Erectile Dysfunction after Nerve-Sparing Radical Retropubic Prostatectomy. Mol Urol. 1999;3(2):109-115. PMID 10851312
- [Background] Berookhim BM, Nelson CJ, Kunzel B, Mulhall JP, Narus JB. Prospective analysis of penile length changes after radical prostatectomy. BJU Int. 2014 May;113(5b):E131-6. doi: 10.1111/bju.12443. Epub 2013 Dec 2. PMID 24053766
- [Background] Kwon YS, Farber N, Yu JW, Rhee K, Han C, Ney P, Hong JH, Lee P, Gupta N, Kim WJ, Kim IY. Longitudinal recovery patterns of penile length and the underexplored benefit of long-term phosphodiesterase-5 inhibitor use after radical prostatectomy. BMC Urol. 2018 May 9;18(1):37. doi: 10.1186/s12894-018-0341-8. PMID 29739455
- [Background] Dalkin BL, Christopher BA. Preservation of penile length after radical prostatectomy: early intervention with a vacuum erection device. Int J Impot Res. 2007 Sep-Oct;19(5):501-4. doi: 10.1038/sj.ijir.3901561. Epub 2007 Jul 26. PMID 17657210
- [Background] Vasconcelos JS, Figueiredo RT, Nascimento FL, Damiao R, da Silva EA. The natural history of penile length after radical prostatectomy: a long-term prospective study. Urology. 2012 Dec;80(6):1293-6. doi: 10.1016/j.urology.2012.07.060. Epub 2012 Oct 23. PMID 23102441
- [Background] Kadono Y, Nohara T, Kawaguchi S, Sakamoto J, Makino T, Nakashima K, Iijima M, Shigehara K, Izumi K, Mizokami A. Changes in penile length after radical prostatectomy: effect of neoadjuvant androgen deprivation therapy. Andrology. 2018 Nov;6(6):903-908. doi: 10.1111/andr.12517. Epub 2018 Jul 2. PMID 29968337
- [Background] Briganti A, Fabbri F, Salonia A, Gallina A, Chun FK, Deho F, Zanni G, Suardi N, Karakiewicz PI, Rigatti P, Montorsi F. Preserved postoperative penile size correlates well with maintained erectile function after bilateral nerve-sparing radical retropubic prostatectomy. Eur Urol. 2007 Sep;52(3):702-7. doi: 10.1016/j.eururo.2007.03.050. Epub 2007 Mar 26. PMID 17418936
- [Background] Engel JD, Sutherland DE, Williams SB, Wagner KR. Changes in penile length after robot-assisted laparoscopic radical prostatectomy. J Endourol. 2011 Jan;25(1):65-9. doi: 10.1089/end.2010.0382. Epub 2010 Nov 29. PMID 21114411
- [Background] Brock G, Montorsi F, Costa P, Shah N, Martinez-Jabaloyas JM, Hammerer P, Ludovico GM, Lee JC, Henneges C, Hamidi K, Rossi A, Mulhall J, Buttner H. Effect of Tadalafil Once Daily on Penile Length Loss and Morning Erections in Patients After Bilateral Nerve-sparing Radical Prostatectomy: Results From a Randomized Controlled Trial. Urology. 2015 May;85(5):1090-1096. doi: 10.1016/j.urology.2014.11.058. Epub 2015 Mar 24. PMID 25813656
- [Background] Toussi A, Ziegelmann M, Yang D, Manka M, Frank I, Boorjian SA, Tollefson M, Kohler T, Trost L. Efficacy of a Novel Penile Traction Device in Improving Penile Length and Erectile Function Post Prostatectomy: Results from a Single-Center Randomized, Controlled Trial. J Urol. 2021 Aug;206(2):416-426. doi: 10.1097/JU.0000000000001792. Epub 2021 Jun 1. PMID 34060339
- [Background] Heo JE, Lee JS, Goh HJ, Jang WS, Choi YD. Urethral realignment with maximal urethral length and bladder neck preservation in robot-assisted radical prostatectomy: Urinary continence recovery. PLoS One. 2020 Jan 13;15(1):e0227744. doi: 10.1371/journal.pone.0227744. eCollection 2020. PMID 31929596
- [Background] Song W, Kim CK, Park BK, Jeon HG, Jeong BC, Seo SI, Jeon SS, Choi HY, Lee HM. Impact of preoperative and postoperative membranous urethral length measured by 3 Tesla magnetic resonance imaging on urinary continence recovery after robotic-assisted radical prostatectomy. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):E93-E99. doi: 10.5489/cuaj.4035. Epub 2017 Mar 16. PMID 28360954
- [Background] Wijkstra PJ, Ten Vergert EM, van Altena R, Otten V, Kraan J, Postma DS, Koeter GH. Long term benefits of rehabilitation at home on quality of life and exercise tolerance in patients with chronic obstructive pulmonary disease. Thorax. 1995 Aug;50(8):824-8. doi: 10.1136/thx.50.8.824. PMID 7570431
- [Background] Savoie M, Kim SS, Soloway MS. A prospective study measuring penile length in men treated with radical prostatectomy for prostate cancer. J Urol. 2003 Apr;169(4):1462-4. doi: 10.1097/01.ju.0000053720.93303.33. PMID 12629384
- [Background] de Rooij M, Hamoen EH, Witjes JA, Barentsz JO, Rovers MM. Accuracy of Magnetic Resonance Imaging for Local Staging of Prostate Cancer: A Diagnostic Meta-analysis. Eur Urol. 2016 Aug;70(2):233-45. doi: 10.1016/j.eururo.2015.07.029. Epub 2015 Jul 26. PMID 26215604
- [Background] Vis AN, van der Poel HG, Ruiter AEC, Hu JC, Tewari AK, Rocco B, Patel VR, Razdan S, Nieuwenhuijzen JA. Posterior, Anterior, and Periurethral Surgical Reconstruction of Urinary Continence Mechanisms in Robot-assisted Radical Prostatectomy: A Description and Video Compilation of Commonly Performed Surgical Techniques. Eur Urol. 2019 Dec;76(6):814-822. doi: 10.1016/j.eururo.2018.11.035. Epub 2018 Dec 2. PMID 30514568